CLINICAL TRIAL: NCT00120029
Title: Peer Counseling for Weight Loss in African American Breast Cancer Survivors
Brief Title: Peer Counseling for Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Collaborators: Barbara Ann Karmanos Cancer Institute (Other); University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 057103MP4F; 1P50ES012395 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer
Keywords: weight loss; survivorship; breast ductal lavage; exercise; diet
MeSH Terms: conditions — Breast Neoplasms; Weight Loss; Motor Activity

INTERVENTIONS:
Behavioral: weight loss counseling

SUMMARY:
The efficacy of peer counseling for weight loss maintenance is being tested in obese and overweight African American breast cancer survivors.

DETAILED DESCRIPTION:
Obesity has adverse effects on breast cancer survival and recurrence, and this may be mediated via the insulin resistance that is associated with obesity. This is a matter of exceptional concern for African-American (AA) breast cancer survivors since a greater proportion of AAs than European Americans (EA) are obese, insulin-resistant and diabetic. This proposal seeks to test the effects of weight loss intervention in obese and overweight AA breast cancer survivors (body mass index 25-40 kg/m2, stage I, II, or IIIA cancer, free of recurrence). Subjects (n=100) will be randomized across 3 arms: 1) control; 2) individualized, dietitian-led counseling; and 3) dietitian-led counseling combined with peer counseling using telephone counseling by trained peers who are AA breast cancer survivors successful at weight control. Psychosocial factors that can affect the extent of weight loss achieved will be assessed, including individual, home and community-level factors. Some of these factors may change when weight loss is achieved and will be assessed both before and after intervention. Genetic polymorphisms that have been shown to be associated with increased body weight, insulin resistance, lipid metabolism, and oxidative stress will be determined and related to both baseline and post-intervention anthropometric and biologic measures. This should further help elucidate inter-individual differences in response to weight loss intervention. The possible beneficial effects of weight loss on the health risks associated with obesity will be evaluated with measures of insulin resistance, insulin-like growth factor and lipid levels in blood samples, as well as with blood pressure and anthropometric measures. The effects of weight loss on these measures have been studied in other obese and overweight populations, but there is little data in breast cancer survivors. Finally, we will attempt to determine if beneficial effects of weight loss can be detected in the breast, since this should be related to subsequent breast cancer risk. The breast contralateral to surgery will be subjected to ductal lavage at baseline, 12 and 24 months. The investigators will examine the effects of weight change on markers of oxidative stress in the breast nipple aspirate fluid that is obtained as part of the lavage procedure. Levels of lipid peroxidation are very high in this fluid and have been related to both nuclear atypia and breast cancer risk. The nuclear morphology of epithelial cells obtained by ductal lavage therefore will be quantified as well. Weight loss in obese and overweight AA breast cancer survivors should improve both psychosocial function and biological indicators of health risks.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* African American
* Up to 7 years post breast cancer diagnosis
* Able to keep food records
* Have a telephone
* Stable weight within 5 pounds last 2 months

Exclusion Criteria:

* Breast cancer recurrence
* History of other cancers
* Uncontrolled congestive heart failure
* Untreated hypertension
* Disabling osteoarthritis
* Abusing drugs or alcohol
* Have psychiatric conditions that interfere with counseling

Ages: 18 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-01; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
markers of oxidative stress in blood and breast fluid
markers of cardiovascular health in blood
body fat
fitness

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, PhD, Principal Investigator — University of Michigan
Locations (1):
- Wayne State University, Detroit, Michigan, United States